CLINICAL TRIAL: NCT03690206
Title: A Phase 3, International, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Glepaglutide in Patients With Short Bowel Syndrome (SBS)
Brief Title: Efficacy And Safety Evaluation of Glepaglutide in Treatment of Short Bowel Syndrome (SBS)
Acronym: EASE SBS 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP1848-17111
Record Dates: First submitted 2018-09-17; First posted 2018-10-01 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Glepaglutide SC injections twice weekly (Experimental): Intervention: Glepaglutide
  Interventions: Drug: glepaglutide
- Glepaglutide SC injections once weekly and placebo once weekly (Experimental): Intervention: Glepaglutide
  Interventions: Drug: glepaglutide; Drug: Placebo
- Placebo SC injections twice weekly (Placebo Comparator): Intervention: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glepaglutide — Glucagon-Like Peptide-2 (GLP-2) analog
  Other Names: ZP1848
  Arms: Glepaglutide SC injections once weekly and placebo once weekly; Glepaglutide SC injections twice weekly
Drug: Placebo — Placebo for glepaglutide
  Arms: Glepaglutide SC injections once weekly and placebo once weekly; Placebo SC injections twice weekly

SUMMARY:
The primary objective of the trial is to confirm the efficacy of glepaglutide in reducing parenteral support volume in patients with short bowel syndrome.

Glepaglutide is the International Nonproprietary Name and USAN for ZP1848.

DETAILED DESCRIPTION:
A Phase 3, international, multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of glepaglutide subcutaneous (SC) injections in patients with short bowel syndrome (SBS).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activity.
* Diagnosis of SBS defined as remaining small bowel in continuity of estimated less than 200 cm and considered stable with regard to PS need. No restorative surgery planned in the trial period.
* Requiring PS at least 3 days per week and maintains a stable PS volume for at least 2 weeks.
* In case of remnant colon: documented colonoscopy which does not give rise to any safety concerns.

Exclusion Criteria:

* More than 2 SBS-related or PS-related hospitalizations within 6 months prior to Screening. No SBS-related hospitalizations within 30 days prior to randomization.
* Poorly controlled inflammatory bowel disease that is moderately or severely active or fistula interfering with measurements or examinations required in the trial.
* Bowel obstruction.
* Known radiation enteritis or significant villous atrophy.
* Cardiac disease defined as: decompensated heart failure (New York Heart Association [NYHA] Class III-IV), unstable angina pectoris, and/or myocardial infarction within the last 6 months prior to Screening.
* Clinically significant abnormal ECG.
* Repeated systolic blood pressure measurements > 180 mm Hg.
* Human immunodeficiency virus positive, acute liver disease, or unstable chronic liver disease.
* Any history of colon cancer. History of any other cancers unless disease-free state for at least 5 years.
* Estimated creatinine clearance < 30 mL/min.
* Severe hepatic impairment.
* Use of GLP-1, GLP-2, human growth hormone, somatostatin, or analogs thereof, within 3 months prior to Screening.
* Use of dipeptidyl peptidase (DPP)-4 inhibitors within 3 months prior to Screening.
* Unstable systemic immunosuppressive therapy within 3 months prior to Screening.
* Unstable biological therapy within 6 months prior to Screening.
* Females of childbearing potential, who are pregnant, breast-feeding, intend to become pregnant or are not using highly effective contraceptive methods.
* Previous exposure to glepaglutide.
* Current, or within 30 days prior to Screening, participation in another interventional clinical trial that includes administration of an active compound.
* Any condition or disease or circumstance that in the Investigator's opinion would put the patient at any undue risk, prevent completion of the trial, or interfere with the analysis of the trial results.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Zealand Pharma
Locations (29):
- United States (7):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Children's Hospital, Chicago, Illinois
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Nashville, Tennessee
- UZ Leuven, Leuven, Belgium
- Canada (3):
  - The Royal Alexandra Hospital, Edmonton
  - Western University, London
  - University Health Network - Toronto General Hospital, Toronto
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- France (2):
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Frankfurt - Med. Klinik I, Frankfurt
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsmedizin Rostock, Rostock
- UMC Radboud Nijmegen, Nijmegen, Netherlands
- Poland (3):
  - Wojewodzki Specjalistyczny Szpital im. M. Pirogowa w Lodzi, Lodz
  - Solumed, Poznan
  - Szpital Skawina sp. z o.o. im. Stanley Dudricka, Skawina
- United Kingdom (5):
  - St Mark's Hospital, Harrow
  - UCLH Foundation NHS Trust, London
  - Salford Royal NHS Foundation Trust, Manchester
  - University of East Anglia, Norwich
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeppesen PB, Vanuytsel T, Subramanian S, Joly F, Wanten G, Lamprecht G, Kunecki M, Rahman F, Nielsen TSS, Berner-Hansen M, Pape UF, Mercer DF. Glepaglutide, a Long-Acting Glucagon-like Peptide-2 Analogue, Reduces Parenteral Support in Patients With Short Bowel Syndrome: A Phase 3 Randomized Controlled Trial. Gastroenterology. 2025 Apr;168(4):701-713.e6. doi: 10.1053/j.gastro.2024.11.023. Epub 2024 Dec 19. PMID 39708985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in (number of sites that randomized patients in parenthesis) Belgium (1), Denmark (2), France (2), Germany (5), the Netherlands (1), Poland (3), Canada (3), the US (7), and the UK (5).
Pre-assignment Details: Patients were diagnosed with SBS and required PS at least 3 days/week. They were willing to adhere to an individual pre-defined drinking menu during 48 h measurement periods and maintain a stable weight.
  The drinking menu and the PS volume and content were adjusted during an optimization phase following by a stabilization phase.
Period: Overall Study
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Started | 35 | 35 | 36
Completed | 31 | 35 | 36
Not Completed | 4 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — ICF withdrawal | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly | Total
Number analyzed (Participants) | 35 | 35 | 36 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 28 | 30 | 81
  >=65 years | 12 | 7 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.4) | 54.0 (12.0) | 55.0 (11.8) | 55.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 20 | 57
  Male | 16 | 17 | 16 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 30 | 33 | 32 | 95
  Unknown or Not Reported | 5 | 1 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 28 | 31 | 30 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 3 | 4
  Netherlands | 2 | 0 | 2 | 4
  Belgium | 3 | 4 | 3 | 10
  United States | 4 | 13 | 6 | 23
  Denmark | 5 | 2 | 1 | 8
  Poland | 8 | 7 | 12 | 27
  United Kingdom | 4 | 4 | 1 | 9
  France | 5 | 1 | 3 | 9
  Germany | 3 | 4 | 5 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.57 (3.35) | 22.72 (3.21) | 23.54 (3.57) | 23.28 (3.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Parenteral Support (PS) Volume
Description: Change in weekly PS volume from baseline to Week 24. Baseline actual weekly PS volume was defined as the actual PS volume derived from a valid 7-day period prior to visit 1 (Day 1), i.e. during the stabilization phase. The actual weekly PS volume at Weeks 1, 2, 4, 8, 12, 16, 20, and 24 was derived as the actual weekly PS volume received during the valid 7-day period prior to the visit. The source for the derivation was the PS volumes recorded by the patients in the eDiary.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one dose of trial drug (glepaglutide or placebo). All efficacy analyses were based on the FAS. Patients were included in the analyses as randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/week
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
L/week | -5.13 [-6.24 to -4.02] | -3.76 [-4.96 to -2.56] | -2.85 [-3.93 to -1.77]
Statistical Analysis 1: Comparison: Glepaglutide SC Injections Twice Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.0039, Mixed Models Analysis; Difference to Placebo = -2.28, 95% CI 2-sided [-3.83 to -0.73]
Statistical Analysis 2: Comparison: Glepaglutide SC Injections Once Weekly and Placebo Once Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.2700, Mixed Models Analysis; Difference to Placebo = -0.91, 95% CI 2-sided [-2.52 to 0.71]

2. Secondary Outcome: Clinical Response in PS Volume
Description: Clinical response, defined as at least 20% reduction in actual weekly PS volume from baseline to both Weeks 20 and 24.
Time Frame: 20 and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 23 | 16 | 14
Statistical Analysis 1: Comparison: Glepaglutide SC Injections Twice Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.0243, Cochran-Mantel-Haenszel; Difference to Placebo = 26.6, 95% CI 2-sided [4.3 to 48.9]
Statistical Analysis 2: Comparison: Glepaglutide SC Injections Once Weekly and Placebo Once Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.6255, Cochran-Mantel-Haenszel; Difference to Placebo = 5.5, 95% CI 2-sided [-16.2 to 27.1]

3. Secondary Outcome: Days Off PS
Description: Achieving 1 or more days per week off PS
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 18 | 12 | 7
Statistical Analysis 1: Comparison: Glepaglutide SC Injections Twice Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel; Difference to Placebo = 31.7, 95% CI 2-sided [11.4 to 51.9]
Statistical Analysis 2: Comparison: Glepaglutide SC Injections Once Weekly and Placebo Once Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.1675, Cochran-Mantel-Haenszel; Difference to Placebo = 13.3, 95% CI 2-sided [-5.4 to 32.0]

4. Secondary Outcome: Clinical Response in PS Volume
Description: Reduction of at least 20 percent in PS volume from baseline to both 12 and 24 weeks.
Time Frame: 12 and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 19 | 15 | 13

5. Secondary Outcome: Weaned Off PS
Description: Reduction in weekly PS volume of 100 percent (weaned off)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 5 | 4 | 0
Statistical Analysis 1: Comparison: Glepaglutide SC Injections Twice Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.0160, Cochran-Mantel-Haenszel; Difference to Placebo = 14.1, 95% CI 2-sided [2.5 to 25.6]
Statistical Analysis 2: Comparison: Glepaglutide SC Injections Once Weekly and Placebo Once Weekly vs Placebo SC Injections Twice Weekly; Test type: Superiority; p = 0.0424, Cochran-Mantel-Haenszel; Difference to Placebo = 11.2, 95% CI 2-sided [0.7 to 21.6]

6. Secondary Outcome: Energy Content
Description: Change in weekly energy content of PS from baseline
Time Frame: 24 weeks
Measure: Median (Full Range); unit: kJ/week
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 26 | 28 | 27
kJ/week | -7360.6 [-48521 to 130351] | -3085.9 [-56550 to 1423] | -734.2 [-46307 to 1670]

7. Secondary Outcome: Days on PS
Description: Change in number of days on PS per week from baseline
Time Frame: 24 weeks
Measure: Median (Full Range); unit: days/week
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 31 | 35 | 36
days/week | -1.00 [-5.0 to 0.0] | 0.00 [-7.0 to 1.0] | 0.00 [-4.0 to 0.0]

8. Secondary Outcome: Change in PS Volume Per Week
Description: Achieving reduction of at least 40 percent in PS volume from baseline to both 20 and 24 weeks
Time Frame: 20 and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 15 | 10 | 8

9. Secondary Outcome: Patient Global Impression of Change Scale (PGIC)
Description: Patient Global Impression of Change scale (PGIC) improvement at Weeks 4, 12, 20, and 24 PGIC improvement was defined as responding "Very Much Improved" or "Much Improved" on a 7-point Likert Scale. Improvement between each glepaglutide treatment regimen compared to placebo was tested by week, using the CMH test adjusted for the stratification factor. Improvement between each glepaglutide treatment regimen versus placebo was tested using collapsed categories of Improvement, No Change, and Worsening, where Improvement is defined as a response of "Very Much Improved" or "Much Improved" or "Minimally Improved", and No Change is defined as the response of "No Change", and Worsening is defined as a response of "Minimally Worse" or "Much Worse" or "Very Much Worse". Improvement using collapsed categories between each glepaglutide treatment regimen compared to placebo was tested by week using a Mantel-Haenszel chi-squared test for ordered categories.
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- Glepaglutide SC Injections Twice Weekly: Intervention: Glepaglutide glepaglutide: Glucagon-Like Peptide-2 (GLP-2) analog
- Glepaglutide SC Injections Once Weekly and Placebo Once Weekly: Intervention: Glepaglutide glepaglutide: Glucagon-Like Peptide-2 (GLP-2) analog Placebo: Placebo for glepaglutide
- Placebo SC Injections Twice Weekly: Intervention: Placebo Placebo: Placebo for glepaglutide
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
participants
  PGIC improved | 22 | 27 | 13
  PGIC much/very much improved | 17 | 11 | 2

10. Secondary Outcome: Safety - Adverse Events
Description: Incidence and type of Adverse Events over an average of 28 weeks (24 weeks treatment + 4 weeks follow up)
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants
  All AEs | 33 | 33 | 27
  Serious adverse events | 9 | 10 | 7
  AE Severity: Severe | 10 | 5 | 2
  AE Severity: Moderate | 15 | 18 | 14
  AE Severity: Mild | 28 | 32 | 24
  Relationship: Related | 27 | 26 | 14
  Relationship: Unlikely related | 18 | 16 | 9
  Relationship: Not related | 26 | 26 | 23
  AEs leading to trial withdrarwal | 2 | 0 | 0
  AEs with action taken drug withdrawn | 2 | 1 | 0
  AEs with action taken drug interrupted | 3 | 0 | 3
  Outcome: Recovered/resolved | 32 | 30 | 25
  Outcome: Recovering/resolving | 7 | 9 | 5
  Outcome: Recovered/resolved with sequelae | 1 | 1 | 0
  Outcome: Not recovered/not resolved | 17 | 14 | 9
  Outcome: Fatal | 0 | 0 | 0
  Outcome: Unknown | 1 | 0 | 0
  Outcome: MIssing | 0 | 0 | 0

11. Secondary Outcome: Number of Patients With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG)
Description: Number of patients with clinically significant changes in ECG will be reported. Monitored ECG parameters included heart rate (beats/min), PR interval (ms), PR interval Aggregate (ms), QRS duration aggregate (ms), QT interval aggregate (ms), QTcF interval aggregate (ms), and RR interval (ms), as well as the overall interpretation of each subject's ECG recorded as Normal, Abnormal Not Clinically Significant, or Abnormal Clinically Significant.
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants | 0 | 0 | 0

12. Secondary Outcome: Safety - Changes in Blood Pressure From Baseline
Description: Changes in blood pressure are reported at Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24 The data collected data are of seated diastolic and systolic blood pressure (mmHg). During treatment phase visits, vital signs were collected before investigational product injection.
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: At certain visits those data are missing for some patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
mmHg
  Week 1 Systolic blood pressure: number analyzed (Participants) | 33 | 30 | 35
  Week 1 Systolic blood pressure | -2.8 [-7.6 to 2.0] | 0.3 [-4.1 to 4.7] | -4.5 [-8.2 to -0.7]
  Week 2 Systolic blood pressure: number analyzed (Participants) | 34 | 30 | 35
  Week 2 Systolic blood pressure | 1.0 [-3.2 to 5.1] | -0.1 [-4.6 to 4.4] | -2.7 [-6.4 to 1.0]
  Week 4 Systolic blood pressure: number analyzed (Participants) | 35 | 29 | 33
  Week 4 Systolic blood pressure | -1.7 [-6.5 to 3.1] | -0.2 [-3.9 to 3.4] | -0.3 [-4.6 to 3.9]
  Week 8 Systolic blood pressure: number analyzed (Participants) | 33 | 29 | 33
  Week 8 Systolic blood pressure | 0.3 [-5.4 to 6.0] | -1.5 [-5.9 to 2.9] | -2.5 [-6.9 to 1.8]
  Week 12 Systolic blood pressure: number analyzed (Participants) | 32 | 29 | 34
  Week 12 Systolic blood pressure | -4.4 [-9.6 to 0.8] | 3.3 [-1.0 to 7.6] | -0.4 [-5.0 to 4.1]
  Week 16 Systolic blood pressure: number analyzed (Participants) | 29 | 32 | 33
  Week 16 Systolic blood pressure | 0.1 [-5.6 to 5.8] | 0.4 [-4.7 to 5.5] | -1.1 [-6.3 to 4.1]
  Week 20 Systolic blood pressure: number analyzed (Participants) | 31 | 28 | 31
  Week 20 Systolic blood pressure | 1.3 [-5.8 to 8.3] | 1.2 [-3.6 to 6.0] | -1.0 [-6.2 to 4.3]
  Week 24 Systolic blood pressure: number analyzed (Participants) | 30 | 33 | 35
  Week 24 Systolic blood pressure | -1.0 [-6.2 to 4.1] | -1.1 [-5.6 to 3.4] | -5.9 [-11.0 to -0.8]
  Week 1 Diastolic blood pressure: number analyzed (Participants) | 33 | 30 | 35
  Week 1 Diastolic blood pressure | 0.4 [-2.3 to 3.0] | 0.5 [-2.6 to 3.5] | -2.0 [-4.6 to 0.6]
  Week 2 Diastolic blood pressure: number analyzed (Participants) | 34 | 30 | 35
  Week 2 Diastolic blood pressure | 2.5 [0.2 to 4.7] | -0.7 [-3.1 to 1.7] | -1.7 [-5.0 to 1.6]
  Week 4 Diastolic blood pressure: number analyzed (Participants) | 35 | 29 | 33
  Week 4 Diastolic blood pressure | 0.0 [-2.8 to 2.8] | -0.2 [-2.5 to 2.8] | -1.5 [-4.6 to 1.6]
  Week 8 Diastolic blood pressure: number analyzed (Participants) | 33 | 29 | 33
  Week 8 Diastolic blood pressure | -0.5 [-3.3 to 2.3] | 1.9 [-1.3 to 5.0] | -0.6 [-3.3 to 2.2]
  Week 12 Diastolic blood pressure: number analyzed (Participants) | 32 | 29 | 34
  Week 12 Diastolic blood pressure | -2.8 [-6.7 to 1.2] | 2.0 [-1.0 to 5.1] | 0.9 [-1.8 to 3.6]
  Week 20 Diastolic blood pressure: number analyzed (Participants) | 31 | 28 | 31
  Week 20 Diastolic blood pressure | 2.1 [-1.5 to 5.7] | -0.7 [-3.9 to 2.4] | 0.4 [-3.3 to 4.1]
  Week 24 Diastolic blood pressure: number analyzed (Participants) | 30 | 33 | 35
  Week 24 Diastolic blood pressure | 2.2 [-1.6 to 5.9] | 0.0 [-2.7 to 2.7] | -0.9 [-3.8 to 2.1]

13. Secondary Outcome: Safety - Changes in Body Temperature From Baseline
Description: Changes in body temperature are reported The body temperature (ºC or ºF) was measured according to the site's usual procedure. During treatment phase visits, vital signs were collected before investigational product injection.
Time Frame: 28 weeks
Population: At certain visits those data are missing for some patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: degree C
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
degree C
  Week 1: number analyzed (Participants) | 33 | 30 | 35
  Week 1 | 0.0 [-0.1 to 0.2] | -0.0 [-0.2 to 0.1] | 0.1 [-0.0 to 0.2]
  Week 2: number analyzed (Participants) | 34 | 32 | 35
  Week 2 | 0.1 [-0.0 to 0.2] | -0.0 [-0.2 to 0.1] | 0.0 [-0.1 to 0.1]
  Week 4: number analyzed (Participants) | 35 | 30 | 33
  Week 4 | -0.1 [-0.2 to 0.1] | -0.0 [-0.2 to 0.1] | 0.1 [-0.1 to 0.2]
  Week 8: number analyzed (Participants) | 33 | 30 | 33
  Week 8 | 0.0 [-0.1 to 0.2] | 0.1 [-0.0 to 0.2] | -0.1 [-0.2 to 0.1]
  Week 12: number analyzed (Participants) | 32 | 29 | 33
  Week 12 | -0.0 [-0.2 to 0.1] | -0.0 [-0.1 to 0.1] | 0.1 [-0.1 to 0.2]
  Week 16: number analyzed (Participants) | 29 | 32 | 34
  Week 16 | -0.0 [-0.1 to 0.1] | -0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1]
  Week 20: number analyzed (Participants) | 31 | 28 | 31
  Week 20 | 0.1 [-0.1 to 0.2] | 0.0 [-0.1 to 0.1] | 0.1 [-0.1 to 0.2]
  Week 24: number analyzed (Participants) | 30 | 33 | 35
  Week 24 | -0.0 [-0.1 to 0.1] | 0.1 [-0.0 to 0.2] | 0.1 [0.0 to 0.2]

14. Secondary Outcome: Immunogenicity - Occurrence of Anti-drug Antibodies
Description: Occurrence of antibodies against glepaglutide The occurrence of glepaglutide-binding antibodies (ADA), M2 binding antibodies (M2 BAb), glepaglutide neutralizing antibodies (NAb) and GLP-2 cross-reacting antibodies (GLP-2 CR) was tested.
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
Number analyzed (Participants) | 35 | 35 | 36
Participants
  ADA (Treatment-induced) | 30 | 31 | 0
  M2 BAb (Treatment-induced) | 28 | 29 | 0
  NAb M2 (Treatment-induced) | 10 | 14 | 0
  GLP-2 CR (Treatment-induced) | 6 | 11 | 0

ADVERSE EVENTS:
Time Frame: All AEs, whether serious or non-serious, were to be reported from the time a signed and dated Informed Consent Form (ICF) was obtained until the end of the post-treatment follow-up period on average 28 weeks.
Description: Due to the long half-life of glepaglutide, all AEs with an onset after the first dose of glepaglutide were treated as 'treatment-emergent', including AEs with an onset during a treatment interruption.
  For the 'Stoma complications' and related preferred terms, the denominators used in the calculation of % are based on patients with small intestine stoma (Glepa 10 mg TW: N=17; Glepa 10 mg OW: N=20; Placebo: N=21).
Arm/Group | Glepaglutide SC Injections Twice Weekly | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly | Placebo SC Injections Twice Weekly
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 9/35 | 10/35 | 7/36
Other Adverse Events (participants affected / at risk) | 30/35 | 31/35 | 25/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Glepaglutide SC Injections Twice Weekly (N=35) | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly (N=35) | Placebo SC Injections Twice Weekly (N=36)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1/17 (1) | 0/20 (0) | 0/21 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Catheter site necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 2 (3) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Glepaglutide SC Injections Twice Weekly (N=35) | Glepaglutide SC Injections Once Weekly and Placebo Once Weekly (N=35) | Placebo SC Injections Twice Weekly (N=36)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Stoma site oedema (Injury, poisoning and procedural complications) | 4/17 (4) | 2/20 (11) | 0/21 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1/17 (1) | 2/20 (2) | 0/21 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 1/17 (1) | 0/20 (0) | 0/21 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Stoma site irritation (Injury, poisoning and procedural complications) | 0/17 (0) | 1/20 (1) | 0/21 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0/17 (0) | 1/20 (1) | 0/21 (0)
Stoma site reaction (Injury, poisoning and procedural complications) | 0/17 (0) | 1/20 (1) | 0/21 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (3) | 3 (7)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 9 (135) | 15 (116) | 1 (1)
Injection site erythema (General disorders) | 5 (6) | 6 (60) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 1 (2)
Fatigue (General disorders) | 4 (4) | 4 (6) | 0 (0)
Injection site pain (General disorders) | 4 (31) | 3 (29) | 0 (0)
Injection site induration (General disorders) | 4 (44) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0) | 2 (2)
Injection site irritation (General disorders) | 3 (13) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 2 (4) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (3) | 4 (22) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 3 (3) | 1 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5) | 6 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03690206/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03690206/SAP_002.pdf